CLINICAL TRIAL: NCT04477421
Title: Femtosecond Small Incision Lenticular Extraction in Comparison to Femtosecond Laser Insitu Keratomileusis Regarding Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Rasheed University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AR200106
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FS-LASIK Group (Active Comparator): 100 eyes of 50 patients underwent bilateral FS-LASIK (Femtosecond laser Insitu Keratomileusis)
  Interventions: Procedure: S-LASIK
- FS-SMILE (Experimental): 100 eyes of 50 patients who underwent bilateral FS-SMILE (femtosecond small incision lenticule extraction)
  Interventions: Procedure: FS-SMILE

INTERVENTIONS:
Procedure: FS-SMILE — Femtosecond small incision lenticule extraction
  Arms: FS-SMILE
Procedure: S-LASIK — Femtosecond laser Insitu keratomileusis
  Arms: FS-LASIK Group

SUMMARY:
Comparison of femtosecond small incision lenticule extraction (FS-SMILE) versus Femtosecond laser Insitu Keratomileusis (FS-LASIK) regarding dry eye disease (DED) and corneal sensitivity (CS) after those refractive surgeries.

ELIGIBILITY:
Inclusion Criteria:

* bilateral eyes with spherical correction range from -2 to -6 diopters and cylinder range from 0 to - 3.5 diopters

Exclusion Criteria:

* sign or symptom of dry eye disease (tear film breakup time (TBUT) >10 seconds
* Schirmer I test >10 mm /5 minutes)
* corneal or conjunctival staining
* Meibomian gland dysfunction
* Previous ocular and or eyelid medical or surgical treatment
* pregnancy
* Chronic systemic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index | After 1 month of surgery
  Ocular Surface Disease Index (the index range from 0 to 100), higher value indicate more severe disease
Ocular Surface Disease Index | After 6 months of surgery
  Ocular Surface Disease Index (the index range from 0 to 100), higher value indicate more severe disease
Tear Break-Up Time | After 1 month of surgery
  Tear Break-Up Time (in seconds)
Tear Break-Up Time | After 6 months of surgery
  Tear Break-Up Time (in seconds)
Schirmer I test | After 1 month of surgery
  Schirmer I test (in mm/5 minutes)
Schirmer I test | After 6 months of surgery
  Schirmer I test (in mm/5 minutes)
Oxford score | After 1 month of surgery
  Oxford score (the score range from 0 to 5), higher value indicate more severe disease
Oxford score | After 6 months of surgery
  Oxford score (the score range from 0 to 5), higher value indicate more severe disease
Dry Eye Work Shop scale | After 1 month of surgery
  Dry Eye Work Shop scale (value range from 0 to 4), higher value indicate more severe disease
Dry Eye Work Shop scale | After 6 months of surgery
  Dry Eye Work Shop scale (value range from 0 to 4), higher value indicate more severe disease

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Rasheed University College, Baghdad, AL-Adhmia, Iraq

IPD SHARING:
Plan to Share IPD: Undecided